CLINICAL TRIAL: NCT05322486
Title: Palliative Primary Tumor Resection in Minimally Symptomatic Patients With Colorectal Cancer and Synchronous Unresectable Metastases Versus Chemotherapy Alone
Brief Title: Palliative Primary Tumor Resection in Minimally Symptomatic Patients With Colorectal Cancer and Synchronous Unresectable Metastases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: State Scientific Centre of Coloproctology, Russian Federation (Other Government)
Responsible Party: Sponsor
Other Study IDs: 22A/20
Record Dates: First submitted 2022-04-02; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Neoplasms, Second Primary; Neoplasm Metastasis; Digestive System Diseases; Gastrointestinal Diseases; Colonic Disease; Intestinal Diseases; Rectal Diseases
Keywords: Colorectal cancer; Primary tumor resection; Minimally symptomatic primary tumor; Unresectable metastases; Chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Neoplasms, Second Primary; Neoplasm Metastasis; Digestive System Diseases; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Rectal Diseases | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary tumour resection group.: Surgical resection of the primary tumour followed by chemotherapy +/- targeted therapy regime.
  Interventions: Procedure: surgery of the primary tumour; Drug: chemotherapy
- Chemotherapy group.: Chemotherapy +/- targeted therapy alone.
  Interventions: Drug: chemotherapy

INTERVENTIONS:
Procedure: surgery of the primary tumour — Surgical resection of the colon tumour, R0. No surgical intervention on metastasis.
  Groups: Primary tumour resection group.
Drug: chemotherapy — Chemotherapy with or without biological drugs.

SUMMARY:
Currently, the question remains whether palliative primary tumor resection could improve overall survival of minimally symptomatic patients with colorectal cancer and synchronous unresectable metastases. The aim of this study is to determine if there is an improvement in overall survival of palliative primary tumor resection followed by chemotherapy in minimally symptomatic patients with colorectal cancer and synchronous unresectable metastases compared to those of upfront chemotherapy/radiotherapy alone.

DETAILED DESCRIPTION:
The present study is a single-center retrospective observational cohort study with a propensity score matching. Between 2016 and 2022 from our institutional database minimally symptomatic patients with colorectal cancer and synchronous unresectable metastases will be selected. Patients will be divided into two groups:

1. Surgical resection of the primary tumour before to systemic therapy
2. Systemic therapy without previous resection of the primary tumour. Propensity score matching (PSM) will be performed, to minimize the selection bias by adjusting variables that may affect the survival of patients. Categorical variables will be compared using the chi-square test or Fisher's exact test. Continuous variables will be compared using the Student's t-test or Mann-Whitney U test. Survival rate will be determined by using Kaplan-Meier analysis with a log-rank test. Univariate and multivariate analyses for survival will be conducted using Cox proportional hazard models. Statistical results will be considered significant at p values less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed colorectal adenocarcinoma
2. Resectable minimally symptomatic primary tumor with unresectable synchronous metastasis
3. Age ≥ 18 years
4. Informed consent

Exclusion Criteria:

1. Synchronous cancers
2. Carcinomatosis
3. Prior surgery, chemotherapy, radiation therapy for the primary tumor or distant metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed with colorectal cancer and synchronous unresectable metastases between 2016 and 2022 from our institutional database.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-29 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 years

SECONDARY OUTCOMES:
Thirty-day mortality | 30 days
Rate of surgical intervention due to complication of treatment | 1 year
Progression free survival (PFS) | 3 years
  PFS is defined as the time interval between the date of diagnosis and the first date of progression of the metastatic disease or death in both treatment arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Ryzhikh National Medical Research Center of Coloproctology, Moscow, Russia